CLINICAL TRIAL: NCT00628602
Title: BION Active Seating for Pressure Ulcer Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Gerald E. Loeb, M.D., Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT8
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Pressure Ulcer
Keywords: Neuromuscular stimulator; Pressure ulcer prevention
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rx Group (Experimental): BION Therapy Group
  Interventions: Device: BION
- Control Group (Placebo Comparator): control group
  Interventions: Device: BION

INTERVENTIONS:
Device: BION — 30 patients operated will be randomized into 2 equal groups, a BION Therapy Group ("Rx group") and a Control Group ("Control group").

SUMMARY:
Pressure ulcers (PUs) are a debilitating pathology resulting from pressure and shear in the soft tissues of immobilized patients. In studies to date, BION neuromuscular stimulation has been demonstrated to activate strong muscle contractions and to produce skeletal motion, with associated increases in muscle bulk (hypertrophy), strength, and metabolic capacity, hence counteracting the 3 major etiological factors in PU development (immobility, soft-tissue atrophy and hypoxia).

This study intends to use neuromuscular stimulation to both shift paralyzed subjects' weight and build up gluteal muscle volume, in order to prevent recurrence of pressure ulcers. We will implant BIONs alongside the already exposed inferior gluteal and sciatic nerves in patients who are undergoing gluteal rotation flap surgery for PU reconstruction. The gluteal rotation flap is a common reconstructive technique for treating PUs by bringing healthy muscle and skin in to repair the deficient area, and to provide healthy tissue covering over bony prominences. The implanted BIONs will enable us subsequently to stimulate the gluteus maximus and hip extensor muscles. Outcome measures will include tissue health variables (measured by clinical assessment, X-Rays, MRI and Sesta-MIBI SPECT perfusion scans), pressure redistribution (measured by an array of pressure sensors), and recurrence rates over 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has had a spinal cord injury and has bilateral lower limb paralysis.
2. Subject cannot contract his/her gluteus muscle voluntarily.
3. Subject is between 18 and 70 years old.
4. Subject sits in a wheelchair for at least 5 hours per day.
5. Attending physician considers the subject in general good health (other than SCI and PU wound).
6. Subject has one or more PUs of Stage III or IV (according to National Pressure Ulcer Advisory Panel Staging1).
7. Subject is having a musculocutaneous (not cutaneous or fasciocutaneous) gluteal rotation flap surgery for PU treatment in which the inferior gluteal pedicle and sciatic nerve will be exposed but not damaged or sacrificed in any way (for any PU wound(s)).
8. Subject is mentally capable of understanding the goals and the application of therapy.
9. Subject is able to apply the therapy (with or without help) once discharged from Rancho Los Amigos.
10. Subject is willing and capable of giving informed consent.
11. Subject is willing and capable of traveling to testing center at the schedules.

Exclusion Criteria:

1. Subject has a positive pregnancy test, is nursing / lactating, or is planning on becoming pregnant or is unwilling to not become pregnant in the next 12 months.
2. Subject has an electronic implant (e.g. cardiac pacemaker, etc.).
3. Subject has any condition associated with a wound healing abnormality (e.g.: connective tissue disorder, immune disorder, diabetes, clinical obesity).

   IDE application: BION Active Seating for Pressure Ulcer Prevention Page 65
4. Subject is malnourished.
5. The attending physician has concerns about the healing of this subject (e.g.: heavy smoking, excessive and/or poorly-managed incontinence).
6. Subject has concurrent concomitant condition affecting the buttock/pelvic area, including other pressure wound not corrected by the flap surgery.
7. Subject suffers from claustrophobia or fear of MRI, or has any contraindication to MRI (e.g. metal implants, pacemaker, etc. not suited to MRI).
8. Subject has damage to the inferior or superior gluteal neurovascular pedicles.
9. Subject is / plans to participate in another investigational study that may affect the healing of PUs or prevent their occurrence/recurrence.
10. Subject is using medications / undergoing procedures that will interfere with NMES effecting muscle contraction (e.g. treatments for spasticity and / or spasms, such as: neurotomies, tenotomies, myotomies, and rhizotomies; as well as tranquilizers and muscle relaxant / paralyzing agents such as Baclofen (Lioresal®), Dantrolene (Dantrium®) and Botulinum Toxin Type A (Botox®)).
11. Subjects whose ulcer extends more than 2.25" deep to the projected surface contour of the buttock when the patient is in a prone position (measured perpendicular to the base of the PU, from the deepest point of the PU to the level of the highest point of the buttock surface, when prone)
12. Subject's wheelchair and the BION system have been tested for interference of either with the other's operation, and either does not operate normally when used together, and this cannot be resolved with an available alternate wheelchair.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Clinical assessment of movement and shifting of weight during BAS. Record shifts in pressure distribution over seated pressure points during NMES. | upon discharge and at the 12-week, 20-week, 36-week and 52-week outpatient follow-up visits.

SECONDARY OUTCOMES:
Clinical Examination of Braden Scale assessment,Reperfusion time,Recurrence of wounds and Body Mass Index | preoperation, upon removal of sutures, upon discharge, and at the 12-week, 20-week, 36-week and 52-week outpatient follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Lucinda Baker, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- Rancho Los Amigos National Rehabilitation Center, Downey, California, United States